CLINICAL TRIAL: NCT01471236
Title: Evaluation of the Agili-C Bi-phasic Implant Performances in the Repair of Cartilage and Osteochondral Defects
Brief Title: Evaluation of the Agili-C Biphasic Implant in the Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0002
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2020-02

CONDITIONS: Cartilage Diseases; Osteochondritis Dissecans
Keywords: cartilage; bone
MeSH Terms: conditions — Cartilage Diseases; Osteochondritis Dissecans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Agili-c bi-phasic implant (Experimental): mini-arthrotomy
  Interventions: Device: Agili-C Bi-phasic Implant; Procedure: mini-arthrotomy

INTERVENTIONS:
Device: Agili-C Bi-phasic Implant — The implantation site should be created in perpendicular manner to the articular cartilage. The surrounding tissue will be cleaned and scraped to prepare a clean site. The implant will be placed in the correct orientation (drilled channels pointing towards the joint side and chamfer towards the bone).
  The implant will be inserted gently in a pressed fit manner.
  Other Names: Agili-C implant
Procedure: mini-arthrotomy — The procedure will be conducted according to hospital practice. The implants will be positioned via open incision, depending on lesion location, and Investigator's final decision. Related treatments during the procedure should be recorded.
  Device positioning details medications and adverse events during the procedure will be recorded. MOCART (off-site), X-ray evaluation (off-site), ICRS Cartilage injury mapping system, Articular cartilage injury Classification and the Osteochondritis Dissecans classification will be recorded.

SUMMARY:
The purpose of this study is to determine the performance of the Agili-C implants. The study hypothesis is that Agili-C implants are effective in the treatment of focal cartilage and cartilage-bone joint surface defects.

DETAILED DESCRIPTION:
Agili-C implant is a bi-phasic, porous resorbable tissue regeneration scaffold for the treatment of focal articular cartilage and for osteochondral defects. Up to 50 patients are to be included in the study. Patients suffering from isolated, single and focal cartilage or osteochondral defect at the knee joint are considered for study inclusion.

ELIGIBILITY:
Inclusion Criteria

1. 18 to 55 years
2. Symptomatic, single, focal, full or near full-thickness (ICRS cartilage defect description grades 3 and 4) chondral or osteochondral isolated lesion of the femoral condyle, trochlea or the tibial plateau

   * Defect area is less than 2 cm² after debridement. The defect is completely surrounded on all sides by healthy cartilage.
   * Osteochondral defect ICRS Cartilage defect description type 1, 2, 3, 4A. Maximal defect depth should be up to 3 millimeters.
3. Primary or secondary articular cartilage repair.
4. Knee is stable or can be stabilized as a concomitant procedure.
5. Must be physically and mentally willing and able to comply with post-operative rehabilitation and routinely schedule clinical and radiographic visits.
6. Signed informed consent.
7. Any misalignments should be fully corrected at the end of the operative procedure.

Exclusion Criteria

1. Uncorrected axial misalignments >5° that cannot be corrected.
2. Patellar cartilage defects or pathology.
3. Meniscal resection of more than 50%, either in a previous procedure or concomitant with articular cartilage repair.
4. Any tumor of the ipsilateral knee, any concurrent malignant tumor or any metastatic tumor in the past or in the present.
5. Active acute or chronic infection of the treated knee.
6. Inflammatory arthropathy or crystal-deposition arthropathy.
7. Systemic cartilage and/or bone disorder; This implants integration is dependent on surrounding live bleeding bone; therefore it must not be implanted within sequestrated or necrotic bone.
8. Bony defect depth over 3 millimeters.
9. Body mass index >35.
10. Asymptomatic articular cartilage defects.
11. Bipolar articular cartilage defects.
12. Osteoarthritis of the operated knee.
13. Oral medications such as systemic corticosteroid therapy taken less than one year prior to surgery or chemotherapy.

    * Previous operative treatment of Arthroscopic marrow stimulation technique or cell therapy operated within the last 6 months
    * Any previous operation of cartilage treatment within the last 6 months
14. Patients who are sensitive to materials containing calcium carbonate or hyaluronate
15. Pregnant women, women who plan to become pregnant and breastfeeding women.
16. Evidence of any significant systemic disease (such as but not limited to HIV infection, hepatitis infection or HTLV infection), known coagulopathies, severe vascular or neurological disease or acute injury that might compromise the patient's welfare.
17. Substance abuse or alcohol abuse.
18. Participation in another clinical trials in parallel to this study.
19. Type I diabetes.
20. Unable to undergo MRI or X-ray.
21. Any reasons making the patient a poor candidate in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
improvement in KOOS pain subscales | 24 months
  The primary efficacy endpoint for this trial will be the change from baseline up to 24 months visit in pain score as measured by the KOOS pain subscale

SECONDARY OUTCOMES:
KOOS total score | 24 months
  * Change from baseline to 3, 6, 9, 12, 18 and 24 months visits as measured by the KOOS total score and subscales.
  * Change from baseline to 18 and 24 months visit in IKDC current health assessment.
  * Change from baseline to 3, 6, 12, 18 and 24 months visit in Lysholm with Tegner knee score.
  * Change from baseline to 3, 6, 12 , 18 and 24 months visit in IKDC knee examination form 2000
  * Change from baseline to 3, 6, 12 , 18 and 24 months visit in IKDC subjective knee evaluation
  * Change in MOCART scoring as measured at 3, 6, 12 , 18 and 24 months visit

OTHER OUTCOMES:
number of SAE | 24 months
  Complications and adverse events, device-related or not, will be evaluated over the course of the clinical trial, including subsequent surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, MD, Principal Investigator
Locations (9):
- Clinical Hospital ''Sveti Duh'', Zagreb, Croatia
- Fakultní nemocnice Brno, Brno, Czechia
- Uzsoki Street Hospital, Budapest, Hungary
- Rizzoli Orthopaedic Institute, Bologna, Italy
- Avimed Hospital, Katowice, Poland
- County Hospital of Timisoara,, Timișoara, Romania
- Serbia (2):
  - Institut Za Ortopediju "Banjica", Belgrade
  - Clinical center of Vojvodina, Novi Sad
- University Medical Centre, Ljubljana, Ljubljana, Slovenia